CLINICAL TRIAL: NCT01182129
Title: Nicotine Delivery and Subjective Effects of 4 mg Nicotine Polacrilex Chewing Gum Compared With Swedish Portion Snus
Brief Title: 4 mg Nicotine Polacrilex Gum and Swedish Portion Snus
Acronym: SMWS06
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Contract Research Organization el AB (Industry)
Collaborators: Swedish Match AB (Industry)
Responsible Party: Erik Lunell, MD, PhD, CROel AB, Slottsvagen 21, SE25284 Helsingborg, Sweden
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SMWS06
Record Dates: First submitted 2010-08-11; First posted 2010-08-16 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy Subjects; Smokers
Keywords: Nicotine Polacrilex chewing gum versus Swedish Snus
MeSH Terms: interventions — Nicotine; Nicotine Chewing Gum; Chewing Gum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Swedish Snus Type 1 (Active Comparator): The subject keeps one pouch of snus still between the upper lip and the gum for 30 minutes. Amount of nicotine extracted, plasma nicotine concentration at 30 minutes (C30), Tmax, Cmax, AUCinf and heart rate for each treatment.
  Interventions: Drug: Nicotine
- Swedish Snus Type 2 (Active Comparator): The subject keeps one pouch of snus still between the upper lip and the gum for 30 minutes. Amount of nicotine extracted, plasma nicotine concentration at 30 minutes (C30), Tmax, Cmax, AUCinf and heart rate for each treatment.
  Interventions: Drug: Nicotine
- 4 mg Nicorette chewing gum (Active Comparator): Nicorette is chewed according to instructions in package insert over 30 minutes.
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Nicotine pouch, 2.2 mg, single dose, 30 minutes
  Other Names: General Onyx 1 g portion snus; General White 1g portion snus
  Arms: Swedish Snus Type 1; Swedish Snus Type 2
Drug: Nicotine — Chewing Gum, 4 mg, single dose, 30 minutes
  Other Names: Nicorette 4 mg chewing gum
  Arms: 4 mg Nicorette chewing gum

SUMMARY:
Fifteen healthy smokers are given single doses of General Onyx 1 g portion snus and General White 1g portion snus, respectively, and one piece of Nicorette 4 mg chewing gum. Serial blood samples are drawn before (0), 2, 4, 8, 16, 24, 30, 45, 60 minutes, 1.5, 2, 4, 6 and 8 hours after administration for determination of nicotine. Mean + SD extracted dose of nicotine from each preparation will be estimated. The percentage extracted of the nicotine content will be calculated. Cmax and Tmax will be estimated. A comparison to Nicorette 4 mg chewing gum will be made. The dose absorbed into the systemic blood circulation (AUC) in relation to the dose following the 4 mg Nicorette chewing gum will be calculated. Self-reports of subjective effects will be obtained up to 30 minutes after the test product is administered using a 100 mm visual analogue scale (VAS) anchored with "not at all" to "extremely". Study hypothesis is that Cmax and AUC of Nicorette 4 mg chewing gum and Swedish snus are similar.

DETAILED DESCRIPTION:
Fifteen healthy smokers are given single doses of General Onyx 1 g portion snus and General White 1g portion snus, respectively, and one piece of Nicorette 4 mg chewing gum. Serial blood samples are drawn before (0), 2, 4, 8, 16, 24, 30, 45, 60 minutes, 1.5, 2, 4, 6 and 8 hours after administration for determination of nicotine. Mean + SD extracted dose of nicotine from each preparation will be estimated. The percentage extracted of the nicotine content will be calculated. Cmax and Tmax will be estimated. A comparison to Nicorette 4 mg chewing gum will be made. The dose absorbed into the systemic blood circulation (AUC) in relation to the dose following the 4 mg Nicorette chewing gum will be calculated. Self-reports of subjective effects will be obtained up to 30 minutes after the test product is administered using a 100 mm visual analogue scale (VAS) anchored with "not at all" to "extremely".

The subjects are male and female smokers, smoking a minimum of 7 cigarettes per day. They should have no history of cardiac, kidney or hepatic disease, alcohol abuse or drug dependence. A physical examination including ECG and blood pressure should give no evidence of disease. No abnormalities should be found in a routine laboratory screening.

The subjects are requested not to smoke or to use any other form of nicotine containing products from 8 p.m. the day before each session until the last blood sample in each session. Previous experience has shown that subjects that have abstained from smoking for 12 hours have a plasma nicotine value of <4 ng/ml. A value >4 ng/ml prior to start of administration should lead to exclusion from statistical analysis. The subjects must be fasting overnight from 12 p.m. the day before each session. No food and drink are allowed from 15 minutes prior to and until 60 minutes after drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer, smoking >7 cigarettes per day. No use of smokeless tobacco and nicotine containing products is allowed. Fasting overnight.

Exclusion Criteria:

* Use of smokeless tobacco and nicotine containing products is not allowed from 8 p.m. the day before trial day. Subjects tested with Smokelyzer for exhaled carbon monoxide.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2006-03; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic/Dynamic Equvivalence | 8 hrs
  After baseline measurements, plasma nicotine concentrations are monitored over 8 hours. Each subject's rating of subjective symptoms, e.g. product "strength" using a 100 mm visual analogue scale (VAS) anchored with "not at all" to "extremely" is recorded up to 30 minutes after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Lunell, MD, PhD, Principal Investigator — Croel AB
Locations (1):
- Carema AB, Eslöv, Skåne County, Sweden